CLINICAL TRIAL: NCT00873925
Title: Transfusion of Autologous Umbilical Cord Blood Plus Vitamin D and Omega 3 Fatty Acids to Preserve Beta Cell Function in Children With Recent Onset Type 1 Diabetes - A Pilot Study
Brief Title: Cord Blood Plus Vitamin D and Omega 3s in T1D
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF IRB 696-2008
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous UCB Plus Vit D Omega 3 FA (Experimental): A single autologous (self) intravenous umbilical cord blood infusion followed by 1 year of daily Vitamin D and Omega 3 Fatty Acid supplementation give as liquid drops and gel capsules that can be swallowed or added to food
  Interventions: Biological: Autologous UCB; Dietary Supplement: Omega 3 FA; Dietary Supplement: Vitamin D
- Control (No Intervention): Subjects randomized to be controls will continue to use intensive insulin therapy in order to compare c-peptide production at 1 year in those receiving combination therapy vs those who do not

INTERVENTIONS:
Biological: Autologous UCB — Umbilical Cord Blood stem cells CAN be collected and frozen immediately after birth in private and public cord blood banks. If a child with recent onset T1D has their OWN cord blood in storage they may qualify for this study. The cells would be released to the University of Florida where we would perform a single IV infusion of the cells once they have been thawed and washed. Depending on how the cells are stored, it may be possible to keep some portion of the cells in storage for future use.
  Arms: Autologous UCB Plus Vit D Omega 3 FA
Dietary Supplement: Omega 3 FA — Omega 3 Fatty Acids commonly found in fish oil may play an important role in preserving beta cell function via their anti-inflammatory actions. Those subjects randomized to treatment will take a daily supplement supplied as a capsule that can either be swallowed whole or opened so the contents can be mixed with food.
  Arms: Autologous UCB Plus Vit D Omega 3 FA
Dietary Supplement: Vitamin D — Vitamin D is important for calcium absorption and bone health but may also play an important role in promoting healthy immune responses. Subjects randomized to intervention will take vitamin D supplied as a liquid in a dropper (1 drop per day added to food) for 1 year.
  Arms: Autologous UCB Plus Vit D Omega 3 FA

SUMMARY:
In this pilot study the investigators are trying to see if a single intravenous infusion of autologous (self) cord blood cells followed by 1 year of daily vitamin D and omega 3 fatty acid supplementation can preserve beta cell function (prolong "honeymoon") in children with type 1 diabetes. All subjects will continue to use insulin therapy as needed to maintain the best possible glucose control.

15 Subjects will be randomized such that 2 of every 3 (10 total) will receive cord blood plus vitamin D and Omega 3 while 1 of 3 (5 total) will serve as controls and will not receive cord blood, vitamin D, or Omega 3 supplementation.

The study will involve 5 visits over 1 year to the University of Florida

This study is a follow-up to our initial study of cord blood infusion alone in which 23 children received autologous cord blood. The initial study was 100% safe but additional studies like the one described above are needed to determine how to improve cord blood based therapy.

DETAILED DESCRIPTION:
Hypothesis: We hypothesize that the combination of intensive insulin therapy, autologous umbilical cord blood (UCB), Vitamin D, and Omega 3 fatty acids administered to children with T1D will preserve residual c-peptide when compared to children receiving intensive insulin therapy alone

Specific Aims:

1. Randomize 15 children with recent onset T1D and available autologous cord blood such that 10 receive a combination of intensive insulin therapy, autologous UCB infusion, and daily Vitamin D while 5 receive intensive insulin therapy alone
2. Document safety of combination therapy
3. Study potential changes in glucose metabolism
4. Study potential changes in immune function

Preliminary Studies: Our group has already performed autologous cord blood infusion in 23 children with T1D and has documented the safety of this approach. While conclusive data regarding the efficacy of the infusion in preserving beta cell function are lacking, our pilot study has demonstrated a potential for cord blood to low the rate of c-peptide decline (a measure of beta cell function/mass) in these young children with T1D. As documented above, considerable work both here and other institutions suggests the potential for a combination of Vitamin D and DHA to further augment the autoimmune response. Given the safety and potential efficacy of such an approach, we feel that a pilot study of the combination of UCB infusion, vitamin D supplementation, and DHA supplementation is warranted.

Screening: Only subjects who are still making at least a small amount of detectable insulin will be eligible for this study. To determine if a child is still making insulin, they will undergo a mixed meal tolerance test. This involves placing an IV in the morning prior to eating. The subject then drinks a "mixed meal" (the nutritional supplement Boost is used)and blood is taken via the IV at timepoints over the next 2 hours to determine if insulin is still being produced.

Randomization: If a potential subject "passes" the screening test, they will then be randomized to either receiving the study intervention or to being a control. Subjects WILL be told what arm of the study they are randomized to.

Infusion: Those randomized to infusion will return to the University of Florida for a single autologous cord blood infusion and will be given vitamin D and Omega 3 supplements

Follow-up: Both Control and Intervention subjects will return at 3, 6, and 12 months after the infusion/screening visit to have blood drawn for a repeat mixed meal tolerance test, measurement of HbA1c, and other immune studies.

ELIGIBILITY:
Inclusion Criteria:

* TID diagnosis confirmed by presence of at least 1 diabetes autoantibody Children ≥ 1 years
* Stored autologous umbilical cord blood (15 sought) in an AABB and/or FACT accredited cord bank.
* Stimulated C-peptide > 0.2pmol/L on MMTT
* Cord blood meets all selection and testing criteria (see below).
* Normal screening values for CBC, Renal function and electrolytes (BMP with Ca, Mg, and Phos).
* Willing to comply with intensive diabetes management

Exclusion Criteria:

* Complicating medical issues that would interfere with blood drawing or monitoring.
* Chronic use of steroids or other immunosuppressive agents for other conditions.
* Positive infectious disease markers from mother's blood or cord at time of -collection (See below for details).
* Any evidence of illness on planned infusion date (i.e. fever >38.5 C, vomiting, diarrhea, wheezing, or crackles).
* Allergy to DHA (Omega 3) or Vitamin D
* Hypercalcemia

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2009-03; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
C-Peptide following the 1 year mixed meal tolerance test | 1 year post cord blood infusion

SECONDARY OUTCOMES:
DHA Level | 1 year post randomization
Vitamin D Level | 1 year post randomization
HbA1c and Insulin Dose | 1 year post randomization
Peripheral Blood T-cell assays | 1 year post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Haller, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Haller MJ, Viener HL, Wasserfall C, Brusko T, Atkinson MA, Schatz DA. Autologous umbilical cord blood infusion for type 1 diabetes. Exp Hematol. 2008 Jun;36(6):710-5. doi: 10.1016/j.exphem.2008.01.009. Epub 2008 Mar 20. PMID 18358588
- [Derived] Haller MJ, Wasserfall CH, Hulme MA, Cintron M, Brusko TM, McGrail KM, Wingard JR, Theriaque DW, Shuster JJ, Ferguson RJ, Kozuch M, Clare-Salzler M, Atkinson MA, Schatz DA. Autologous umbilical cord blood infusion followed by oral docosahexaenoic acid and vitamin D supplementation for C-peptide preservation in children with Type 1 diabetes. Biol Blood Marrow Transplant. 2013 Jul;19(7):1126-9. doi: 10.1016/j.bbmt.2013.04.011. Epub 2013 Apr 20. PMID 23611977